CLINICAL TRIAL: NCT00765440
Title: Role of Peri-operative Immunonutrition in Cancers of the Higher Aero-digestive Tract
Brief Title: Study of Nutrition Regimens in Treating Patients With Cancer of the Upper Aerodigestive Tract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2006/26; 2007-A00091-52 (Other: AFSSAPS ID RCP)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2015-02

CONDITIONS: Head and Neck Cancer; Infection; Malnutrition
Keywords: infection; malnutrition; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Infections; Malnutrition; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (Placebo Comparator): Patients receive standard oral or enteral nutrition (IMPACT® placebo) over 7 days prior to surgery and over 7 days after surgery.
  Interventions: Other: placebo
- Arm II (Experimental): Patients receive oral or enteral neoadjuvant IMPACT® nutrition over 7 days prior to surgery and enteral adjuvant standard nutrition (IMPACT® placebo) over 7 days after surgery.
  Interventions: Dietary Supplement: therapeutic nutritional supplementation; Other: placebo
- Arm III (Experimental): Patients receive oral or enteral IMPACT® nutrition over 7 days prior to surgery and enteral adjuvant IMPACT® nutrition over 7 days after surgery.
  Interventions: Dietary Supplement: therapeutic nutritional supplementation

INTERVENTIONS:
Dietary Supplement: therapeutic nutritional supplementation — Given orally
  Arms: Arm II; Arm III
Other: placebo — Given orally
  Arms: Arm I; Arm II

SUMMARY:
RATIONALE: It is not yet known which regimen of enteral nutrition is more effective in preventing infections in patients undergoing surgery for cancer of the upper aerodigestive tract.

PURPOSE: This randomized phase III trial is comparing three nutrition regimens in treating patients with cancer of the upper aerodigestive tract.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of immunonutrition (IMPACT®) in patients with de novo cancer of the upper aerodigestive tract.

Secondary

* Determine the best time to initiate treatment.
* Compare the intermediate duration of treatment.
* Compare nutritional parameters.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive standard oral or enteral nutrition (IMPACT® placebo) over 7 days prior to surgery and over 7 days after surgery.
* Arm II: Patients receive oral or enteral neoadjuvant IMPACT® nutrition over 7 days prior to surgery and enteral adjuvant standard nutrition (IMPACT® placebo) over 7 days after surgery.
* Arm III: Patients receive oral or enteral IMPACT® nutrition over 7 days prior to surgery and enteral adjuvant IMPACT® nutrition over 7 days after surgery.

After completion of study therapy, patients are followed at 30 days after surgery and then at 2 and 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of de novo cancer of the upper aerodigestive tract, including the following:

  * Oral cavity
  * Larynx
  * Oropharynx
  * Hypopharynx
* Planned surgical excision of tumors with opening of the mucous membranes, with or without immediate reconstruction by myocutaneous pedicle flap or free-bone graft
* Planned adjuvant enteral nutritional regimen lasting at least 7 days post-operatively

PATIENT CHARACTERISTICS:

* ANC > 1.8 x 10^9/L
* Hemoglobin > 9 g/dL
* Transaminases ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 3 times ULN
* Creatinine 70-250 μmol/L
* Urea ≤ 1.5 times ULN
* Glucose < 1.5 g/L
* Sodium < 145 mmol/L
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No psychological, social, geographical, or familial reasons prohibiting follow-up
* No insulin-dependent diabetes
* No severe psychiatric illness

PRIOR CONCURRENT THERAPY:

* No head and neck surgery for cancer within the past year
* No prior oral components of immunonutrition
* No prior neoadjuvant chemotherapy
* No prior radiotherapy to head and neck

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rate of infectious complication | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noelle Falewee Pastor, Study Chair — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- [Derived] Falewee MN, Schilf A, Boufflers E, Cartier C, Bachmann P, Pressoir M, Banal A, Michel C, Ettaiche M. Reduced infections with perioperative immunonutrition in head and neck cancer: exploratory results of a multicenter, prospective, randomized, double-blind study. Clin Nutr. 2014 Oct;33(5):776-84. doi: 10.1016/j.clnu.2013.10.006. Epub 2013 Oct 17. PMID 24182765